CLINICAL TRIAL: NCT00778856
Title: Hand Transplantation for the Reconstruction of Below the Elbow Amputations
Acronym: VCA-01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator relocated to another institution
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Linda C Cendales, MD, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007760
Record Dates: First submitted 2008-10-07; First posted 2008-10-24 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Amputation; Transplantation
MeSH Terms: interventions — Hand Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand Transplant (Experimental)
  Interventions: Procedure: Hand transplantation

INTERVENTIONS:
Procedure: Hand transplantation — allotransplantation of deceased donor composite tissue (hand and forearm)

SUMMARY:
Organ transplantation has become the treatment of choice for most patients suffering end stage diseases of the kidney, pancreas, liver, heart or lung.

Vascularized Composite Allotransplantation (VCA) {a.k.a. composite tissue allotransplantation} is the term used to describe transplantation of multiple tissues (skin, muscle, bone, cartilage, nerve, tendon, vessel) as a functional unit (e.g. hand). Several recent advances in clinical organ transplant immunosuppression and experimental limb VCA have now made it feasible to consider clinical VCA for the functional restoration of patients with loss of one or both hands.

This protocol facilitates the development of limb VCA at the Atlanta Veterans Affairs Medical Center (VAMC) and at Emory University for patients with below the elbow amputations. It will evaluate the patients' use of transplanted limb(s) in activities of daily living and compare the function of the transplanted hand to the function with their previous prosthesis.

Patients with below the elbow amputations will be enrolled. Donor tissue will be recovered from deceased donors following the guidelines of and in cooperation with the regional Organ Procurement Organization. The transplantation procedure and postoperative care will be performed using the standard technique for limb replantation. Patients will receive standard immunosuppressive regimen. Rejections will be treated in keeping with experience from the solid organ transplant experience. Graft failure will be treated with allograft amputation.

DETAILED DESCRIPTION:
This protocol will study patients with below the elbow amputations who are selected to undergo limb allotransplantation. We will study patients after they have been trained on the use of a prosthetic limb device prior to transplantation. We will treat them with immunosuppression known to prevent the rejection of other allografted tissues and designed to minimize their dependence on chronic maintenance immunosuppression. These patients will be studied to determine whether the transplanted limb functions better, worse or the same as a prosthetic hand, and to quantify those differences

ELIGIBILITY:
Inclusion Criteria:

* male or female, 18-55 years of age, with below elbow amputation
* ability to give informed consent

Exclusion Criteria:

* Any condition that precludes serial follow-up.
* Any active malignancy or any history of a hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing these are appropriately eliminated prior to transplant. For amputations due to malignancy, 5 years recurrence free survival will be required prior to enrollment.
* Any known immunodeficiency syndrome.
* Inability or unwillingness to comply with protocol monitoring and therapy, including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services
* Pregnancy or unwillingness to practice birth control methods during the first year of the study.
* Unwillingness to undergo blood transfusion if clinically indicated

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ability-relative to prosthetic limbs-to use the transplanted limb in activities of daily living, measured by quantitative functional tests | 18 months

SECONDARY OUTCOMES:
Incidence of hand allograft rejection | 2 years
Development/presence of alloantibodies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda C. Cendales, MD, Principal Investigator — Emory University School of Medicine, VA Medical Center
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia